CLINICAL TRIAL: NCT04825288
Title: A Phase I/II Randomized, Double-blind, Placebo-controlled Trial (1-BETTER) Examining XB2001 (Anti-IL-1⍺ True Human Antibody) in Combination With ONIVYDE + 5-FU/LV (+Folinic Acid) in Advanced Pancreatic Cancer
Brief Title: XB2001 in Combination With ONIVYDE + 5-FU/LV (+Folinic Acid) in Advanced Pancreatic Cancer
Acronym: 1-BETTER
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: XBiotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-PT049
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects in phase II portion will be randomized on a 1:1 basis to XB2001 plus ONIVYDE + LV + 5-FU (Arm 1) or placebo plus ONIVYDE + LV + 5-FU (Arm 2).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): XB2001 + ONIVYDE + 5-FU + LV combination therapy administered for 12 cycles of treatment
  • Arm 1 Treatment Cycle: Patients randomized to this arm will receive the following treatments every 2 weeks: XB2001 MTD as an intravenous infusion over up to 60 minutes, followed by ONIVYDE 70 mg/m2 intravenously over 90 minutes, followed by leucovorin l + d racemic 400 mg/m2 intravenously over 30 minutes, followed by 5-Fluorouracil 2400mg/m2 intravenously over 46 hours. Therapy will be administered every 2 weeks (2 weeks = 1 cycle).
  Interventions: Biological: XB2001 or Placebo
- Arm 2 (Placebo Comparator): Placebo + ONIVYDE + 5-FU + LV combination therapy administered for 12 cycles of treatment
  • Arm 2 Treatment Cycle: Patients randomized to this arm will receive the following treatments every 2 weeks: Placebo as an intravenous infusion over up to 60 minutes, followed by ONIVYDE 70 mg/m2 intravenously over 90 minutes, followed by leucovorin l + d racemic 400 mg/m2 intravenously over 30 minutes, followed by 5-fluorouracil 2400 mg/m2 intravenously over 46 hours. Therapy will be administered every 2 weeks (2 weeks = 1 cycle).
  Interventions: Biological: XB2001 or Placebo

INTERVENTIONS:
Biological: XB2001 or Placebo — XB2001 is a True Human monoclonal antibody that blocks the biological activity of IL-1α with a high degree of affinity and specificity. IL-1⍺ is a key mediator of inflammatory responses and is implicated in the pathophysiology of various diseases, including cancer, cardiovascular and rheumatologic diseases. Ample evidence supports targeting IL-1⍺ to block pathological inflammatory processes associated with many diseases.

SUMMARY:
This trial will include 2 portions (phase 1 and phase 2).

The first portion will be a Phase I, open label, dose escalation study to establish the maximum tolerated dose (MTD) of XB2001 as measured by Dose-Limiting Toxicity (DLT), in combination with ONIVYDE + LV + 5-FU chemotherapy regimen in patients with advanced pancreatic cancer and to determine the recommended dose for the subsequent Phase 2 study.

The phase 2 portion will be implemented with the maximum established tolerated dose (MTD) of XB2001. The target enrollment in the phase 2 portion is 60 patients which will be randomized on a 1:1 basis to XB2001 plus ONIVYDE + LV + 5-FU (Arm 1) or placebo plus ONIVYDE + LV + 5-FU (Arm 2).

DETAILED DESCRIPTION:
Study Title: A Phase I/II randomized, double-blind, placebo-controlled trial (1-BETTER) examining XB2001 (anti-IL-1⍺ True Human antibody) in combination with ONIVYDE + 5-FU/LV (+folinic acid) in advanced pancreatic cancer

Sponsor: XBiotech USA, Inc.

Study Chair: David Park, M.D.

Sample Size: Approximately 69 patients will be enrolled in the USA (at least 9 patients in the open label phase 1 portion and 60 patients in the randomized phase 2 portion)

Approximate Duration:

This trial will include 2 phases. The first portion will be a Phase I, open label, dose escalation study evaluating the safety, tolerability and establishing the Maximum Tolerated Dose (MTD) of XB2001 in at least nine patients with metastatic pancreatic adenocarcinoma who are receiving ONIVYDE + Leucovorin l + d racemic + 5-Fluorouracil chemotherapy treatment. The duration for each patient in the Phase I portion will be 14 days (1 treatment cycle) in which they will be given one intravenous dose of XB2001 prior to receiving ONIVYDE + Leucovorin l + d racemic + 5-Fluorouracil chemotherapy treatment and assessed for Dose Limited Toxicities (DLT). The Phase II portion will be implemented following the completion of the Phase I portion and declaration of the MTD. The duration of subject participation in the randomized, double-blind, placebo-controlled Phase II portion of the trial is approximately 28 weeks: including a screening period of up to 30 days, and 24-week treatment period. All study subjects can continue treatment with XB2001 in an open label extension, for as long as they are judged to be benefitting clinically and have had no unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed pancreatic adenocarcinoma of exocrine pancreas that is metastatic, unresectable, or recurrent
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumor V1.1
* Documented disease progression after one prior gemcitabine-based therapy OR one FOLFIRINOX and gemcitabine combination therapy
* Eastern Cooperative Oncology Group (ECOG) performance of 0 or 1 or Karnofsky performance status (KPS) ≥ 70
* Adequate hepatic, renal and bone marrow function

Exclusion Criteria:

* Clinically significant decrease in performance status (medical records) within 2 weeks of intended first dose administration
* Clinically significant GI disorders
* Severe arterial thromboembolic events less than 6 months before inclusion
* Prior Whole Brain Radiation Therapy (WBRT)
* Evidence of brain metastases
* NYHA Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure (defined as ≥ 160/100 mm Hg)
* Use of strong CYP3A4 inducers or inhibitors and/or UGT1A1 inhibitors within 14 days prior to Visit 1/Baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD) of XB2001 as measured by Dose-Limiting Toxicity (DLT), in combination with ONIVYDE + LV + 5-FU chemotherapy regimen in patients with advanced pancreatic cancer. | 44 days
  Primary Endpoint for Phase I portion
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | 28 weeks
  Safety endpoints will be evaluated for number of subjects by monitoring treatment emergent adverse events (TEAE) from clinical and laboratory reporting as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Progression Free Survival | From baseline until the date of first documented disease progression or date of death (from any cause), whichever come first, assessed up to 24 weeks.
  Progression Free Survival will be evaluated following the formal database lock, or during an interim analysis, if applicable. PFS is defined as the time from date of randomization to the date of disease progression or death (any cause). Disease progression can include clinical progression, in which it is deemed by the investigator that the patient is coming off study due to the progression of underlying disease. Clinical or radiological (RECIST 1.1) progression will suffice as disease progression.
Overall Survival (OS) | From baseline until the date of death (from any cause) assessed up to 24 weeks.
  Overall survival (OS) will be defined as the duration from the date of randomization until death. Subjects who are alive at the end of follow-up will be censored and survival time will be defined as time from randomization to censor date.
Objective Response Rate | Assessment every 8 weeks after initial response assessed up to 24 weeks.
  Objective Response Rate will be defined by the percent of patients in the study with a best overall response of CR or PR as assessed by the investigator (per RECIST 1.1).
Time to Treatment Failure | From baseline to treatment discontinuation (any cause) assessed up to 24 weeks
  Time to treatment failure is defined as a composite endpoint measuring time from randomization to discontinuation of treatment for any reason, including disease progression, treatment toxicity, or death.
Percentage of Patients with Clinical Benefit Response | Baseline to weeks 8, 16 and 24. CBR will be defined as a composite measure consisting of change in lean body mass (LBM) and change in quality of life
  For Phase 2 portion only. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. The CBR will be defined as a stabilization or positive (≥0 kg) change in lean body mass (LBM)-as assessed by dual-energy X-ray absorptiometry (DEXA) scan, and improvement or no worsening (≥0 score point change) on any two of the three symptom scale measures (fatigue, pain, appetite) of EORTC QLQ-C30
Quality of Life assessed through the cancer-specific European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life questionnaire (QLQ)-C30 | Baseline to weeks 8, 16 and 24
  Score ranges from 0 to 100. A high score represents a higher response level.
Number of Serious Adverse Events (SAEs) | From baseline (Visit 1) (post-infusion) until two weeks after the last infusion, assessed up to 24 weeks
  For Phase 2 portion only
Incidence of Grade 3-4 Diarrhea | From Visit 1 (post-infusion) until two weeks after the last infusion, assessed up to 24 weeks
  For Phase 2 portion only
Duration of hospitalizations | Baseline to weeks 4, 8, 12, 16, 20 and 24
  For Phase 2 portion only
Plasma/serum concentration of XB2001 | At the specified timepoints in the study calendar assessed up to 24 weeks
  Plasma/serum concentration of XB2001 will be measured throughout the study.
Number of Treatment Cycles | Throughout the study assessed up to 24 weeks
  For Phase 2 portion only
Change in (CD14+CD16+IL-1⍺+) triple positive tumor associated monocytes in peripheral blood | Baseline to week 2 (post infusion at visit 2)
  For Phase 2 portion only

OTHER OUTCOMES:
Results of a symptom questionnaire will be summarized by treatment arm at various post-infusion time points and compared over time | At various post-infusion time points assessed up to 22 weeks
  Score ranges from 12 to 48. A high score represents worse outcome.
Cardiotoxicity measured by the number of required ECGs and cardiotoxicity related events summarized by treatment arm and compared over time | Compared over time, assessed up to 22 weeks
  Exploratory Endpoint (Phase 2 portion only)

CONTACTS AND LOCATIONS:
Overall Officials: David J Park, Study Chair — Providence St. Joseph Heritage
Locations (28):
- United States (28):
  - Arizona Oncology Associates, Tucson, Arizona
  - Disney Family Cancer Center at Providence St. Joseph Medical Center, Burbank, California
  - TOI Clinical Research, Cerritos, California
  - Providence St. Joseph Heritage - Fullerton, CA, Fullerton, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Sarah Cannon - Florida Cancer Specialists, Lake Mary, Florida
  - Mt. Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Alliance for Multispecialty Research, LLC, Merriam, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Revive Research - Farmington Hills, Farmington Hills, Michigan
  - Revive Research - Sterling Heights, Sterling Heights, Michigan
  - St. Vincent Frontier Cancer Center, Billings, Montana
  - Summit Medical Group, Florham Park, New Jersey
  - Stony Brook Cancer Center, Stony Brook, New York
  - Montefiore Einstein Medical Center, The Bronx, New York
  - Providence Portland, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center Cancer Institute, Knoxville, Tennessee
  - Sarah Cannon - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Bon Secours St. Francis Cancer Center, Midlothian, Virginia

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available